CLINICAL TRIAL: NCT01543126
Title: A Prospective Study Assessing the Correlation Between Disease Prognosis and the Level of IL-6 and IL-8 Level in Blood and Pleural Effusion Before and After Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: IL-6 and IL-8 Level of Blood and Pleural Effusion During Chemotherapy in Metastatic Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: it's too slow to enroll suitable patients into this study
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Principal Investigator, Fudan University
Other Study IDs: Fudan BR2011-06
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pleural effusion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pleural effusion: patients with pleural effusion

SUMMARY:
Change of IL-6 and IL-8 level in blood and pleural effusion before and after chemotherapy correlate with the prognosis of the disease

DETAILED DESCRIPTION:
To assess the correlation between the disease prognosis and the level of IL-6 and IL-8 in blood and pleural effusion before and after chemotherapy in patients with metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 70 years old;
* Patients with histologic proved metastatic breast cancer;
* Pleural effusion with the volume of more than 1000ml, as documented by CT, X ray or ultrasound;
* There are no other diseases which cause the elevation of IL-6 or IL-8, such as cirrhosis of liver, anaphylactoid purpura, acute pancreatitis;
* With at least one measurable disease according to RECIST criteria,
* Normal laboratory results:ANC≥2.0×109/L,Hb≥80g/L,plt≥100×109/L,TB<UNL (<1.5 x UNL in patients with liver mets),ALT/AST< 1.5 x UNL (<2.5x UNL in patients with liver mets),AKP<5 x UNL(except bone mets),Cr<UNL;
* Normal functions with heart, liver,renal and bone marrow;
* Got ICF before enrollment;
* Life expectancy more than 12 weeks.

Exclusion Criteria:

* Pregnant or breast-feeding women or positive serum pregnancy test;
* Uncontrolled brain metastases;
* No recovery from previous radiation or accepted radiation within 4 weeks before enrollment;
* Participation in any investigational drug study within 4 weeks preceding treatment start;
* Concurrent other malignancy at other sites or previous other cancer within the last 5 years, with the exception of adequately treated in situ carcinoma of cervix uteri or basal or squamous cell carcinoma of the skin;
* Serious uncontrolled intercurrent infections;
* Poor compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer patients with pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
level of IL-6 and IL-8 | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD.PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China